CLINICAL TRIAL: NCT00002386
Title: A Multiclinic, Open Pilot Study to Investigate the Effect of Combination Antiretroviral Therapy Including Indinavir Sulfate on Coagulation Factors, on Platelet Aggregation, and on Factor VIII/IX Half-Life in HIV-1 Seropositive Patients With Hemophilia A or B
Brief Title: Effect of Indinavir Plus Two Other Anti-HIV Drugs on Blood Clotting in HIV-Positive Males With Hemophilia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 246J; 065-00
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections; Hemophilia A
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Indinavir; Factor VIII; Factor IX; Half-Life; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Platelet Aggregation; Hemophilia A; Hemophilia B
MeSH Terms: conditions — HIV Infections; Hemophilia A; Hemophilia B | interventions — Indinavir; Lamivudine; Stavudine; Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if indinavir plus two other anti-HIV drugs affect blood clotting in HIV-positive patients with hemophilia.

DETAILED DESCRIPTION:
Patients are enrolled in one of two study groups. The treatment group consists of HIV-1 seropositive patients with hemophilia A or B who are protease-inhibitor naive. The laboratory control group consists of HIV-1 seropositive patients with hemophilia A who are on a stable, triple-combination antiretroviral regimen. Patients in the treatment group receive indinavir sulfate plus two of the following NRTIs: zidovudine (ZDV), didanosine (ddI), zalcitabine (ddC), stavudine (d4T), or lamivudine (3TC). Patients in the treatment group preferably are naive to one or both of the NRTIs. Patients in the laboratory control group continue on their stable triple antiretroviral regimen consisting of a protease inhibitor plus two NRTIs. Patients in the control group are not provided antiretroviral medications as part of this study. Patients in the treatment group are evaluated by physical examination, safety laboratory tests, CD4 cell counts, and viral load on Day 1 and at Weeks 2, 4, 8, and 12 and then every 8 weeks through Week 52. Patients in the control group are evaluated by physical examination, safety laboratory tests, CD4 cell counts, and viral load on Day -1 and at Week 12. All patients receive their usual factor concentrate infusion over a 10-minute period on Day -1 and at Week 12 to estimate factor VIII (or IX) recovery and half-life. Blood samples are taken prior to infusion and 30 minutes and 1, 3, 6, 9, 12, and 24 hours after infusion. All patients are required to keep a daily log documenting bleeding episodes and use of factor VIII (or IX) throughout the study.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are an HIV-positive male.
* Have been diagnosed with hemophilia.
* Have been taking clotting factors for hemophilia for at least 6 months.
* Have been taking a combination of one protease inhibitor plus two other anti-HIV drugs for at least 6 months, or have never taken a protease inhibitor.
* Are at least 16 years old (consent of parent or guardian required if under 18).

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - USCF, San Francisco, California
  - Georgetown U Med Ctr / Div of Hematology / Oncology, Washington D.C., District of Columbia
  - Emory Univ, Atlanta, Georgia
  - Riley Hosp for Children, Indianapolis, Indiana
  - Tulane Univ School of Medicine / Hematology / Oncology, New Orleans, Louisiana
  - Univ of North Carolina School of Medicine / Div Hemat / Onco, Chapel Hill, North Carolina
  - Milton Hershey Med Ctr, Hershey, Pennsylvania
- Montreal Gen Hosp, Montreal, Quebec, Canada